CLINICAL TRIAL: NCT01271309
Title: Migratory and Angiogenic Dysfunction of Circulating CD133 Stem Cells: a New Prognostic Marker in Myocardial Ischemia.
Brief Title: Stem Cell Migratory Activity: Prognostic Marker in Myocardial Ischemia
Status: Completed | Type: Observational
Sponsor: IRCCS Multimedica (Other)
Collaborators: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Other Study IDs: 05/2007_Ferrara
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Myocardial Infarction patients: Patients with thoracic pain lasting at least 20 min and ST changes or left B block, not present in previous ECG.

SUMMARY:
The present project aims to determine whether a deficit in migration of stem cells could be implicated in the failure to mount an adequate collateralization after Myocardial Infarction (MI) and thereby facilitate the development of post-ischemic heart failure (HF) and to dissect underlying molecular mechanisms. Furthermore, the investigators wish to determine the predictive value of stem cell migration assay in patients with MI.

DETAILED DESCRIPTION:
MAIN OBJECTIVES OF THE STUDY:

Characterization of circulating CD133+ stem cells in a group of 170 patients with MI (mean post-MI follow up, 6 months):

* Counting total mononuclear cells and FACS analysis of CD133 stem cells.
* Characterization of CD133+ stem cell biology: Migratory assay, imaging of cytoskeleton, angiogenesis tests in vitro.
* Evaluation of migratory signalling, with specific focus on the PI3K/Akt/eNOS system.

Assessment of the prognostic value of the stem cell migration assay.

* Relationship between cell biology tests on CD133+ cells and changes in circulating cytokines and pro-angiogenic factors after MI.
* Assessment of area at risk by ECG-synchronized Single Photon Emission Computed Tomography (gated-SPECT) in subgroups with different patterns of stem cell migratory tests.
* Assessment of ventricular remodelling (echocardiography, NMR) in relation with patterns of stem cell migratory test.

EXPECTED RESULTS:

Clarification of the implication of stem cell migratory deficit in post-ischemic HF.

* Identification of underlying mechanisms
* Identification of a cellular marker for prediction of patients at risk of HF.

RELEVANCE TO PUBLIC HEALTH:

* Introduction of a biological test for the early diagnosis of post-MI HF
* Recognition of therapeutic targets for the rescue of stem cell migratory liabilities

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Thoracic pain lasting at least 20 min and ST changes or left B block, not present in previous ECG.
* MI confirmed by elevation of troponin I and CK-MB.
* Patients with Killip II e III LV dysfunction will be included.

Exclusion Criteria:

* Patients reporting thoracic pain 24 hours prior to hospitalization
* HF symptoms resistant to therapy
* Haemoglobin< 10 gr/dl
* Haemodynamic instability (systolic pressure <90 mmHg after treatment)
* Alterations in haematopoiesys
* Concurrent neoplastic disease
* No written informed consent or other conditions that affect patient's compliance to protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited sequentially at the Operative Unit of Ferrara having the following characteristics: Thoracic pain lasting at least 20 min and ST changes or left B block, not present in previous ECG. MI will be confirmed by elevation of troponin I and CK-MB. Patients will be treated according to international guidelines. With regard to medical treatment, this will include all available drugs except for statins, which will be inserted only 14 days post-MI, to avoid the confounding effect of these drugs on stem cell biology.
  Patients reporting thoracic pain 24 hours prior to hospitalization will be excluded. Similarly, those with HF symptoms resistant to therapy will be excluded. By contrast, patients with Killip II e III LV dysfunction will be included.
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Prognostic value of CD133+ stem cells in MI | 12 months
  Correlation of clinical parameters of disease evolution and biological features

SECONDARY OUTCOMES:
Correlation of disease evolution and other biomarkers | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, MD, Principal Investigator — University Ferrara Hospital
Locations (2):
- Italy (2):
  - Cardiology Dept. Arcispedale S.Anna, Ferrara
  - IRCCS Multimedica, Milan

REFERENCES:
- [Result] Fortunato O, Spinetti G, Specchia C, Cangiano E, Valgimigli M, Madeddu P. Migratory activity of circulating progenitor cells and serum SDF-1alpha predict adverse events in patients with myocardial infarction. Cardiovasc Res. 2013 Nov 1;100(2):192-200. doi: 10.1093/cvr/cvt153. Epub 2013 Jun 12. PMID 23761401